CLINICAL TRIAL: NCT05351424
Title: Audiovisual Didactic Experience for Latinx Patient Treatment Adherence and Non-English Speaker Trial Enrollment (ADELANTE) Study in Radiation Oncology
Brief Title: AVI Didactic Experience for Latinx Patient Treatment Adherence and Non-English Speaker Trial Enrollment Study in Rad Onc
Acronym: ADELANTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Lisa A. Kachnic, Professor and Chair, Department of Radiation Oncology, Columbia University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAT2490
Record Dates: First submitted 2022-03-31; First posted 2022-04-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Invasive; Prostate Cancer
Keywords: breast cancer; prostate cancer; audiovisual intervention; Spanish-speaking; focus group; treatment experience; patient education; radiotherapy adherence; cancer trial participation
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 2x2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Audiovisual Intervention- Radiation Therapy Education (Experimental): Audiovisual video will be provided to the subjects as educational material.
  Interventions: Other: Audiovisual Intervention- Radiation Therapy Education
- Written Brochure- Radiation Therapy Education (Active Comparator): Written brochures will be provided to the subjects as educational material.
  Interventions: Other: ASTRO Radiation Therapy for Breast or Prostate Cancer Brochure
- Audiovisual Intervention- Cancer Clinical Trials (Experimental): Audiovisual video will be provided to the subjects as educational material.
  Interventions: Other: Audiovisual Intervention- Cancer Clinical Trials Education
- Written Brochure- Cancer Clinical Trials (Active Comparator): Written brochures will be provided to the subjects as educational material.
  Interventions: Other: NCI Taking Part in Cancer Research Studies Brochure

INTERVENTIONS:
Other: Audiovisual Intervention- Radiation Therapy Education — A video with educational information will be shown regarding radiation therapy.
  Arms: Audiovisual Intervention- Radiation Therapy Education
Other: ASTRO Radiation Therapy for Breast or Prostate Cancer Brochure — Brochure with written information will be given to the subject regarding radiation therapy.
  Arms: Written Brochure- Radiation Therapy Education
Other: Audiovisual Intervention- Cancer Clinical Trials Education — A video with educational information will be shown regarding cancer clinical trials.
  Arms: Audiovisual Intervention- Cancer Clinical Trials
Other: NCI Taking Part in Cancer Research Studies Brochure — Brochure with written information will be given to the subject regarding cancer clinical trials.
  Arms: Written Brochure- Cancer Clinical Trials

SUMMARY:
The study aims to develop educational media interventions to prepare Latinx Spanish-speaking radiation oncology patients for a course of breast or prostate cancer radiation therapy and to foster receptivity and informed decision-making around cancer clinical trial participation.

DETAILED DESCRIPTION:
Research suggests that utilization of audiovisual educational interventions may help to address health literacy and language barriers as well as suboptimal outcomes and trial enrollment in minority and/or non-English speaking patients. However, this has yet to be demonstrated in the radiation oncology setting, in which educational material is limited to written brochures for non-English speaking patients. Herein, the investigators propose to develop and implement a targeted linguistically and culturally appropriate audiovisual intervention (AVI) for Latinx/Spanish-speaking (SS) patients undergoing curative radiotherapy (RT). Our overall objective is to demonstrate benefit of AVI on RT knowledge, adherence, satisfaction and cancer trial perceptivity and enrollment in Latinx/SS patients. The investigators also aim to identify patient-specific and modifiable system-level factors predictive of quality RT delivery and clinical trial accrual to instruct future demographic-segmentation strategies focused on reducing outcomes disparities within radiation oncology.

ELIGIBILITY:
Pilot Phase Inclusion Criteria:

1. Spanish speakers of Latinx background as defined by the U.S. Census Bureau as anyone from Mexican, Puerto Rican, Cuban, Dominican, Central or South American ancestry
2. Currently undergoing treatment for breast or prostate cancer, or recently been treated

Pilot Phase Exclusion Criteria:

1. Patient with bilateral deafness and/or blindness
2. Patient with psychosis and/or dementia

Main Study Inclusion Criteria:

1. Spanish speakers of Latinx background as defined by the U.S. Census Bureau as anyone from Mexican, Puerto Rican, Cuban, Dominican, Central or South American ancestry
2. Patients with non-metastatic prostate or breast cancer
3. Histopathologically proven diagnosis of prostate or breast cancer
4. History and physical examination within 28 days prior to enrollment
5. Karnofsky performance status 70 or greater
6. For women of childbearing potential, pregnancy testing to be performed in accordance to institutional guidelines
7. Plan to receive definitive, curative radiation. Patients planning to receive curative RT after upcoming adjuvant chemotherapy or induction hormonal therapy may enroll at reconsult "follow-up" visit.
8. Consultation visit must be performed with a certified interpreter

Main Study Exclusion Criteria:

1. Patient with bilateral deafness and/or blindness
2. Patient with psychosis and/or dementia
3. Clinical or radiological evidence of metastatic disease
4. Prior participation in cancer patient education trial
5. Prior RT
6. RT for sites other than breast or prostate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with breast cancer, and males with prostate cancer.
Enrollment: 194 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiation Therapy (RT) Knowledge Questionnaire | : baseline prior to first randomization (within 1 week of enrollment for both breast and prostate cancer) and before CT simulation visit, and again during CT simulation visit (1-4 weeks from enrollment for both breast and prostate cancer)
  Subjects will complete the "RT Knowledge Questionnaire" to measure the change in the subjects' understanding of radiation therapy. This will be administered twice- once prior the subject receiving either the AVI or written brochure on RT knowledge and before CT simulation, and again on the same day after CT simulation.
Radiation Therapy (RT) Adherence Score | up to 6 weeks after completion of Radiation Therapy
  Reflects the frequency of unplanned treatment and clinic absence as well as subject compliance of provider recommendations
Radiation Therapy (RT) Satisfaction Questionnaire | during or immediately prior to the end-of-treatment visit (4-6 weeks from enrollment for breast cancer, 4-9 weeks from enrollment for prostate cancer)
  Adapted for radiation oncology setting from the CAHPS Cancer Center and EORTC Cancer Patient Satisfaction Surveys

SECONDARY OUTCOMES:
Clinical Trials Perceptivity Questionnaire | Prior to second randomization during the last week of radiation therapy (4-6 weeks after enrollment for breast cancer, 4-9 weeks for prostate cancer) and again during the first follow-up visit after completing radiation therapy (8-12 weeks from e
  Subjects will complete the "Clinical Trials Perceptivity Questionnaire" to measure the change in the subjects' understanding of cancer clinical trials. This will be administered twice- once during the last week of RT prior to the subject receiving either the AVI or written brochure on cancer clinical trials, and again during the first follow-up visit after completing radiation therapy.
Clinical trial enrollment | following completion of RT (4-6 weeks from enrollment for breast cancer, 4-9 weeks for prostate cancer), for up to 5 years
  Subjects' medical records will be reviewed to ascertain the number subsequent cancer clinical trials they enroll in after completing radiation therapy, for up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Kachnic, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No